CLINICAL TRIAL: NCT06325566
Title: A Prospective, Multicenter, Randomized, Double-blind, Controlled Study to Evaluate the Efficacy and Safety of a Single Injection of Rexlemestrocel-L Combined With HA in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety of Rexlemestrocel-L Combined With HA* in Participants With Moderate to Severe Chronic Low Back Pain
Acronym: HyaluronicAcid
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSB-DR004
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rexlemestrocel-L + HA (Experimental): Participants will receive rexlemestrocel-L 2.0 mL injection of approximately 6 million rexlemestrocel-L cells in freeze media mixed in a 1:1 by-volume ratio with hyaluronic acid (HA) solution on Day 0.
  Interventions: Drug: Rexlemestrocel-L + HA mixture
- Control Group (Sham Comparator): Participants will receive saline solution as a sham procedure to simulate the active treatment injection on Day 0.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Rexlemestrocel-L + HA mixture — Rexlemestrocel-L will be combined in 1:1 by-volume ratio with HA solution and the resulting mixture will be administered as intradiscal injection.
  Arms: Rexlemestrocel-L + HA
Drug: Saline — Saline solution injection adjacent to the index disc.
  Arms: Control Group

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of rexlemestrocel-L+HA compared to control in reducing low back pain at 12 months post-treatment and safety of a single injection of rexlemestrocel-L+HA injected into a lumbar intervertebral disc compared to control through 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe low back pain for a duration of at least six months who have failed at least 3 months of conservative care.
* Participants who have moderate radiographic degeneration of an intervertebral disc from L1 to S1, with a single disc suspected of causing chronic lower back pain (CLBP).

Exclusion Criteria:

* Participants who have been a recipient of prior allogeneic stem cell/progenitor cell therapy for any indication or autologous stem cell/progenitor cell therapy or other biological intervention to repair the index intervertebral disc.
* Participants with low back pain duration of less than 6 months or greater than 60 months.
* Participants who have not received at least 3 months of conservative treatment for back pain without adequate pain relief.
* Participants taking systemic immunosuppressants.
* Participants with osteoporosis.
* Participants with alcohol or substance abuse problems.
* Participants with severe depression or anxiety.
* Participants with cauda equina syndrome; fibromyalgia, symptomatic central vertebral canal stenosis, lumbar spondylitis or other undifferentiated spondyloarthropathy affecting the index disc.
* Participants having undergone a surgical procedure affecting the structure/biomechanics of the disc (e.g., discectomy, intradiscal electrothermal therapy, intradiscal radiofrequency, artificial disc replacement, interbody fusion, laminectomy, etc.) at the index or adjacent levels.
* Participants who have received any lumbar intradiscal injection into the index disc or adjacent discs within three months prior to the start of screening, other than injection of contrast medium for discography.
* Participants who received an epidural steroid injection within 6 weeks prior to informed consent.
* Participants with evidence of neurologic deficit on any component of the lumbar neurological exam at baseline.
* Participants with sacroiliac (SI) joint pain, as determined by a targeted physical exam, or SI joint injection.
* Participants with facet joint pain, as determined by a medial branch block.
* Participants with more than a single painful level.
* Participants with a full thickness annular tear observed on magnetic resonance imaging (MRI) or discography.
* Participants with low back pain that is less than moderate in severity.
* Participants with extreme low back pain.
* Participants who lack moderate to extreme functional limitations/disability.

Note: Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Daily Average Low Back Pain at 12 Months Post-treatment Based on Visual Analog Scale (VAS) Score | Baseline and Month 12
  Low back pain intensity will be measured using a VAS ranging from 0-100 millimeter (mm). A score of 0 represents no pain and 100 represents worst possible pain.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Month 24

SECONDARY OUTCOMES:
Percentage of 30% VAS Pain Responders at 12 Months Post-treatment | Month 12
  Responders are defined as participants who have at least a 30% decrease from baseline in daily average low back pain VAS score (measured as the average VAS score over 7 days). VAS score ranges from 0 (no pain) to 100 (worst possible pain).
Mean Change From Baseline in Quality of Life Measured by Euroqol-5D (EQ-5D) Index Score at 12 Months Post-treatment | Baseline and Month 12
  The EQ-5D is a generic instrument that consists of 5 dimensions: Mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression, rated over five levels of severity ranging from no issues to extreme issues and the responses can be converted into a single number called an index score. The index scores are calculated ranging from 0 (worst quality of life) to 1 (perfect quality of life).
Percentage of Minimal Pain Responders at 12 Months Post-treatment | Month 12
  Minimal pain responders are defined as participants who have a low back pain daily average VAS score (measured as the average VAS score over 7 days) of 20 mm or less. VAS score ranges from 0 (no pain) to 100 (worst possible pain).
Mean Change From Baseline in Function as Measured by Oswestry Disability Index (ODI) Questionnaire Score at 12 Months Post-treatment | Baseline and Month 12
  ODI scores ten aspects of the participant's home and work life and analgesic use in a range of 0 (least amount of disability) to 5 (severe disability). The disability index is then calculated by summing the scores for all questions answered, then multiplied by two and reported in a 0 to 100% range where higher numbers indicate a higher level of disability.
Percentage of Participants With 30% VAS and 10-point ODI Treatment Success at 12 Months Post-treatment | Month 12
  Treatment success based on the percentage of participants who have at least a 30% reduction from baseline in daily average low back pain VAS score (measured as the average VAS score over 7 days) with at least a 10-point decrease from baseline ODI score will be reported.
Percentage of Participants Who Ceased Opioid Usage at 24 Months Post-treatment | Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Roger D Brown, Study Director — Mesoblast, Ltd.
Locations (39):
- United States (39):
  - Axsendo Clinical Research/Summa Pain Care, Phoenix, Arizona
  - Pain Institute of Southern Arizona, Tucson, Arizona
  - TriWest Research Associates, Chula Vista, California
  - Boomerang Health Care, Concord, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Newport Therapeutics, Newport Beach, California
  - University of California-Davis Spine Center, Sacramento, California
  - Innovative Pain Treatment Solutions, San Diego, California
  - University of California-San Francisco, San Francisco, California
  - Source Healthcare, Santa Monica, California
  - Colorado Spine Partners/The Denver Spine and Pain Institute, Greenwood, Colorado
  - Prime Medical Research, Coral Gables, Florida
  - Cantor Spine Center at the Paley Orthopedic & Spine Institute, Fort Lauderdale, Florida
  - New Life Medical Research Center, Hialeah, Florida
  - Bold City Clinical Research, Jacksonville, Florida
  - OSSO Health, Inc., Miami Beach, Florida
  - Interventional Pain Institute, The Villages, Florida
  - Conquest Research LLC, Winter Park, Florida
  - Emory Healthcare, Dunwoody, Georgia
  - Vista Clinical Research, Newnan, Georgia
  - Hawaii Pain & Spine, Kailua, Hawaii
  - University of Kansas Medical Center, Kansas City, Kansas
  - Iqra Research, Edgewood, Kentucky
  - Paradigm Health System, Slidell, Louisiana
  - The Kahan Center, Annapolis, Maryland
  - Reno Tahoe Pain Associates, Reno, Nevada
  - University of Rochester, Rochester, New York
  - Eximia EquiHealth Research LLC/Emerge Ortho, Durham, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Meta Medical Research Institute, LLC, Dayton, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Axsendo Clinical Research/Compass Pain and Wellness, Portland, Oregon
  - OSS Health, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Paradigm Research Center/Houston Scoliosis and Spine Institute, Houston, Texas
  - Axsendo Clinical Research/Texas Institute of Pain and Spine, Pearland, Texas
  - VA iSpine Physicians, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No